CLINICAL TRIAL: NCT04054245
Title: Open Label Phase 2 Single Agent Study of PAT-1251 in Patients With Primary Myelofibrosis (PMF), Post-Polycythemia Vera Myelofibrosis (Post-PV MF), or Post-Essential Thrombocytosis Myelofibrosis (Post-ET MF)
Brief Title: PAT-1251 in Treating Patients With Primary Myelofibrosis, Post-Polycythemia Vera Myelofibrosis, or Post-Essential Thrombocytosis Myelofibrosis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: "Company is in a process of being taken over by another pharma and the new one has different ideas on how to pursue studies with this drug"
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0831; NCI-2019-03143 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0831 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2019-06-06; First posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Myelofibrosis Transformation in Essential Thrombocythemia; Polycythemia Vera, Post-Polycythemic Myelofibrosis Phase; Primary Myelofibrosis
MeSH Terms: conditions — Polycythemia Vera; Primary Myelofibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (LOXL2 inhibitor PAT-1251) (Experimental): Patients receive LOXL2 inhibitor PAT-1251 PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: LOXL2 Inhibitor PAT-1251; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: LOXL2 Inhibitor PAT-1251 — Given PO
  Other Names: PAT-1251; PAT1251; PAT 1251; Lysyl Oxidase-like Protein 2 Inhibitor PAT-1251
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well PAT-1251 works in treating patients with primary myelofibrosis, post-polycythemia vera myelofibrosis, or post-essential thrombocytosis myelofibrosis. PAT-1251 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy of LOXL2 inhibitor PAT-1251 (PAT-1251) as therapy for primary myelofibrosis (PMF), post-polycythemia vera (PV) myelofibrosis (MF), and post-essential thrombocytosis (ET) MF.

II. To determine the objective response of PAT-1251 treatment which is defined as CR (complete remission) + PR (partial remission) + CI (clinical improvement) after three and six cycles of treatment.

SECONDARY OBJECTIVES:

I. To determine the safety of PAT-1251 as therapy for PMF, post-PV MF and post-ET MF.

II. To determine time to response and response duration. III. To assess changes in symptom burden as assessed by Myeloproliferative Neoplasm Symptom Assessment Form Total Symptom Score (MPN-SAF TSS).

EXPLORATORY OBJECTIVES:

I. To explore changes in bone marrow reticulin fibrosis, collagen, osteosclerosis (grading).

II. To determine the percent target engagement based on a plasma target engagement assay after treatment with PAT-1251.

OUTLINE:

Patients receive LOXL2 inhibitor PAT-1251 orally (PO) twice daily (BID) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must provide written informed consent
* Willing and able to comply with scheduled visits, treatment plan and laboratory tests
* Patient is able to swallow and retain oral medication
* Must be diagnosed with treatment requiring PMF or post ET/PV MF with intermediate -1, intermediate -2 or high risk disease according to the International Working Group (IWG) prognostic scoring system, or if with low risk disease then with symptomatic splenomegaly that is greater than or equal to 5 cm below left costal margin by physical exam
* Patients who are not candidates for, intolerant of, or relapsed/refractory to ruxolitinib
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (1500/mm^3)
* Serum direct bilirubin =< 2.0 x ULN (upper limit of normal)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) or alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) (if both measured, then this applies to both measurements) =< 2.5 x ULN, except for patients with MF involvement of the liver who must have levels =< 5 x ULN
* Treatment-related toxicities from prior therapies must have resolved to grade =< 1
* At least 2 weeks from prior MF-directed treatment (till the start of study drug)

Exclusion Criteria:

* Any concurrent severe and/or uncontrolled medical conditions that could increase the patient's risk for toxicity while in the study or that could confound discrimination between disease- and study treatment-related toxicities
* Impaired cardiac function or clinically significant cardiac diseases, including any of the following:

  * History or presence of ventricular tachyarrhythmia
  * Presence of unstable atrial fibrillation (ventricular response > 100 beats per minute [bpm]); patients with stable atrial fibrillation are eligible, provided they do not meet any of the other cardiac exclusion criteria
  * Clinically significant resting bradycardia (< 50 bpm)
  * Angina pectoris or acute myocardial infarction =< 3 months prior to starting study drug
  * Other clinically significant heart disease (e.g., symptomatic congestive heart failure; uncontrolled arrhythmia or hypertension; history of labile hypertension or poor compliance with an antihypertensive regimen)
* Patients who are currently receiving chronic (> 14 days) treatment with corticosteroids at a dose >= 10 mg of prednisone (or its glucocorticoid equivalent) per day, or any other chronic immunosuppressive treatment that cannot be discontinued prior to starting study drug
* Patients with impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of PAT-1251 as per physicians opinion
* Pregnant or breast feeding (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive - human chorionic gonadotropin (HCG) laboratory test
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 90 days after study treatment. Highly effective contraception methods include:

  * Total abstinence or
  * Male partner or female sterilization or
  * Combination of any two of the following (a+b or a+c, or b+c):

    * Use of oral, injected or implanted hormonal methods of contraception
    * Placement of an intrauterine device (IUD) or intrauterine system (IUS)
    * Barrier methods of contraception: condom for male partner or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository
  * Note: Postmenopausal women are allowed to participate in this study. Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of asomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, a woman is considered to be of not child bearing potential only when her reproductive status has been confirmed by follow-up hormone level assessment
* Sexually active males must use a condom during intercourse while taking the drug and for 3 months after stopping study drug and should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2019-07-24 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 6 cycles, each cycle is 28 days.
  Will be defined as complete remission (CR) + partial remission (PR) + clinical improvement (CI). Responses will be categorized according to the revised International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) and European Leukemia Net (ELN) consensus criteria for myelofibrosis. Will be estimated along with the exact 95% confidence interval.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 2 years
  Toxicity is defined as grade 3-4 clinically relevant non-hematologic toxicity or a serious adverse event that is at least possibly drug related (Common Terminology Criteria for Adverse Events version 4.03) and occurs anytime during the treatment. The method of Thall, Simon and Estey will be used for toxicity monitoring. Safety data will be summarized by category, severity and frequency. The proportion of patients with AEs will be estimated, along with the Bayesian 95% credible intervals.
Time to response | From date of first treatment to the first date at which the subject's objective status was classified as a response (CR, PR, or CI), assessed up to 2 years
  The distribution will be estimated by Kaplan-Meier curves.
Duration of response | From the date at which the patient's objective status is first noted to be a CR, PR, or CI to the date of progression (no longer meeting criteria for either CR, PR, or CI) is documented (if one has occurred), assessed up to 2 years
  The distribution will be estimated by Kaplan-Meier curves.
Changes in symptom burden | Baseline up to 2 years
  Will be assessed by Myeloproliferative Neoplasm Symptom Assessment Form Total Symptom Score.
The Descriptive statistics in the improvement of anemia | Baseline up to 2 years
  Will be used to explore improvements in anemia and the following outcomes will be summarized: mean changes in hemoglobin at monthly intervals.
The Descriptive statistics in Improvements of transfusion dependence. | Baseline up to 2 years
  Will be used to explore improvements in the transfusion dependence. The following outcomes will be summarized: mean changes in hemoglobin at monthly intervals.
The Transfusion of independent patients | Baseline up to 2 years
  Will be summarized if the patient is not requiring transfusions on the study who experience an increase of 2 g/dL in their hemoglobin.
Proportion of transfusion dependent patients who become transfusion independent | Baseline up to 2 years
  The proportion of transfusion dependent patients (defined as requiring a transfusion of 2 units packed red blood cells (PRBCs) monthly for 3 months (12 weeks) prior to starting the trial) who become transfusion independent (not requiring a transfusion of PRBCs over a period of 3 months (12 weeks) while on study) will be summarized.
Proportion of transfusion dependent patients who become transfusion independent and have a 1 g/dL increase in hemoglobin | Baseline up to 2 years
  Will be summarized.
Proportion of transfusion independent patients requiring a transfusion | Baseline up to 2 years
  Will be summarized.

OTHER OUTCOMES:
The Correlative Studies | Baseline up to 2 years
  Descriptive statistics including plots, mean, median and standard deviations will be used to summarize data. For continuous outcomes, t-test and analysis of variance (ANOVA) will be used to compare outcome measures across patient characteristics. Dunnett's and Tukey's test that properly adjust for multiplicity in multiple tests will be implemented. Pair-wise comparisons will be performed using pre- and post-therapy samples from each patient. The chi-square test or Fisher's exact test will be used to test the association between two categorical variables such as disease state and performance status.
Percent target engagement after treatment | Baseline up to 2 years
  The percent target engagement based on a plasma target engagement assay after treatment with LOXL2 inhibitor PAT-1251 will be determined. Descriptive statistics including plots, mean, median and standard deviations will be used to summarize data. For continuous outcomes, t-test and ANOVA will be used to compare outcome measures across patient characteristics. Dunnett's and Tukey's test that properly adjust for multiplicity in multiple tests will be implemented. Pair-wise comparisons will be performed using pre- and post-therapy samples from each patient. The chi-square test or Fisher's exact test will be used to test the association between two categorical variables such as disease state and performance status.

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Masarova, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org